CLINICAL TRIAL: NCT03622424
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study Assessing the Effects of Gelesis200 on Appetite Parameters, Food Intake, and Glycemic Control in Overweight or Obese Subjects With or Without Diabetes: A Sub-Study of LIGHT-UP
Brief Title: Effects of Gelesis200 on Appetite Parameters, Food Intake, and Glycemic Control in Overweight or Obese Prediabetic Subjects: A Sub-Study of LIGHT-UP
Acronym: MATCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gelesis, Inc. (Industry)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GS-200-003
Record Dates: First submitted 2017-09-12; First posted 2018-08-09 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-04

CONDITIONS: Overweight and Obesity; PreDiabetes; Type2 Diabetes
MeSH Terms: conditions — Overweight; Obesity; Prediabetic State

STUDY DESIGN:
Intervention Model Description: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study Assessing the Effects of Gelesis200 on Appetite Parameters, Food Intake, and Glycemic Control in Overweight or Obese Prediabetic Subjects: A Sub-Study of LIGHT-UP
Who Masked: Participant, Care Provider, Investigator
Masking Description: Subjects, investigators, and sponsor will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gelesis200 (Active Comparator): Subjects on this ARM will receive Gelesis200
  Interventions: Device: Gelesis200
- Placebo (Placebo Comparator): Subjects on this ARM will receive a placebo device
  Interventions: Device: Placebo
- Gelesis200 and Placebo (Active Comparator): Subejcts on this ARM will receive both Gelesis200 and placebo.
  Interventions: Device: Gelesis200 and Placebo

INTERVENTIONS:
Device: Gelesis200 — Gelesis200: Three (3)Gelesis200 capsules (2.10 g) three (3) times per day (i.e., breakfast, lunch, and dinner)
  Arms: Gelesis200
Device: Placebo — Placebo: Three (3)placebo capsules three (3) times per day (i.e., breakfast, lunch, and dinner)
  Arms: Placebo
Device: Gelesis200 and Placebo — Placebo and Gelesis200: Three (3) placebo capsules at breakfast,and three (3) Gelesis200 capsules (2.10 g)two (2) times per day (i.e., lunch and dinner)
  Arms: Gelesis200 and Placebo

SUMMARY:
This study evaluates the effects of Gelesis200 on Appetite Parameters, Food Intake, and Glycemic Control in Overweight or Obese Prediabetic Subjects: A Sub-Study of LIGHT-UP. Some of the patients will receive Gelesis200, the other will receive a combination of Gelesis200 and placebo and the final group will receive just placebo.

DETAILED DESCRIPTION:
Overweight (BMI ≥25 and <30kg/M2) and obesity (BMI ≥30kg/M2) are major health problems, world-wide. The overweight/obesity epidemic was first noted in the US and then spread to other industrialized nations, and is now seen even in developing countries. The World Health Organization (WHO) estimated that the worldwide prevalence of obesity has nearly doubled between 1980 and 2008, and in a separate analysis, the NCD Risk Factor Collaboration (NCD RisC) and the WHO estimated that the worldwide prevalence of diabetes has nearly quadrupled between 1980 and 2014, from 108 million to 422 million, respectively.

The intra-gastric balloon is an intervention designed to reduce stomach volume, but there are conflicting data on sustained weight loss and no clear data indicating a decrease in mortality. Side effects include balloon movement, nausea, vomiting, pain, and stomach ulceration. The results from bariatric surgery suggest that limiting the functional volume of the stomach is an effective modality for the treatment of obesity. However, because of the invasive nature of the procedure, associated risk of peri-operative complications and the relatively high cost, bariatric surgery is usually reserved for the severely obese subjects. A need exists for a product that is easy to use, safe, convenient, more accessible, and effective at inducing and sustaining weight loss. Interventions which act mechanically by occupying stomach volume, increasing the elasticity and viscosity of the upper gastrointestinal content, and extending gastric emptying time, could potentially be very beneficial.A medical device which induces satiety and decreases hunger could result in decreased caloric intake and weight loss. The advantage of such a medical device is that it would not require drastic restriction of food choices and would circumvent the challenge of unacceptable hunger levels which have derailed so many dietary interventions in the past.

Gelesis200, when hydrated, is homogeneously mixed with the ingested food,increasing the volume and elasticity of the stomach and small intestine contents. This in turn may induce satiety,which reduces food intake. Previous studies with a similar hydrogel (Gelesis100) have shown increased satiety,reduced body weight(especially in prediabetics), and improved glycemic control. It is expected that Gelesis200 will have similar effects to Gelesis100. Furthermore, the physical properties of Gelesis200 (viscosity), which are similar to some dietary fibers, suggest that Gelesis200 will have a favorable impact on glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ambulatory subjects
* Age ≥22 years and 65 years
* Body Mass Index (BMI) ≥27 and ≤40 kilogram (kg)/meter (M)2 with body weight <120 kg
* Prediabetic subjects with FPG ≥100 milligram (mg)/deciliter (dL) and <126 mg/dL [≥5.6 millimole (mmol)/liter (L) and <7.0 mmol/L] at both Screening Visits with HbA1c ≤6.4% [≤46 mmol/mole (mol)] [if only one (1) value is within this range, the other value should not be ≥126 mg/dL (≥7.0 mmol/L) and HbA1c should be ≥5.7% (≥39 mmol/mol) and ≤6.4% (≤46 mmol/mol)], untreated diabetic subjects with FPG ≤ 200 mg/dL (≤ 11.2 mmol/L) at both Screening Visits and either FPG ≥126 mg/dL (≥7.0 mmol/L) at both Screening Visits or HbA1c ≥6.5% (≥48 mmol/mol) if FPG is <126 mg/dL (<7.0 mmol/L) at one (1) or both Screening Visits, or metformin-treated diabetic subjects with FPG ≥70 mg/dL and ≤270 mg/dL (≥3.9 mmol/L and ≤15.1 mmol/L) at both Screening Visits
* Fasting serum insulin <24 microunit ([Symbol]U)/milliliter (mL) at both Screening Visits in prediabetic subjects
* Ability to follow verbal and written instructions
* Consent obtained via signed ICF

Exclusion Criteria:

* Pregnancy [or positive serum or urine pregnancy test(s) in females of childbearing potential]
* Absence of medically approved contraception in females of childbearing potential [exempli gratia (e.g.), hysterectomy, oral contraceptive medications, intrauterine device combined with a barrier method, two (2) combined barrier methods such as diaphragm and condom or spermicide, or condom and spermicide; bilateral tubal ligation and vasectomy are acceptable contraceptive methods when combined with another single method from above]
* History of allergic reaction to carboxymethylcellulose (CMC), citric acid, maltodextrin, gelatin, or titanium dioxide
* Participation in a weight loss study within the past twelve (12) months
* Administration of Gelesis100 or Gelesis200 in a previous study
* Administration of investigational products within one (1) month prior to Screening Visit
* Smoking cessation within six (6) months prior to Screening Visit or considering smoking cessation during the study
* Anticipated surgical intervention during the study period
* Known Type 1 Diabetes
* History of eating disorders including binge eating (except for mild binge eating) or emesis ≥2/week from any cause
* Weight change >3% within three (3) months prior to and during the Screening period
* Supine systolic blood pressure (SBP) >160 millimeters of mercury (mmHg) and/or supine diastolic blood pressure (DBP) >95 mmHg
* Angina, coronary bypass, or myocardial infarction within six (6) months prior to Screening Visit
* History of swallowing disorders
* Esophageal anatomic abnormalities (e.g., webs, diverticuli, rings)
* History of gastroesophageal reflux disease
* History of gastric or duodenal ulcer
* History of gastroparesis (e.g., chronic nausea, vomiting ≥2 occurrences per week, heartburn, etc.)
* History of gastric bypass or any other gastric surgery
* History of small bowel resection (except if related to appendectomy)
* History of intestinal stricture (e.g., Crohn's disease)
* History of intestinal obstruction or high risk of intestinal obstruction, including suspected small bowel adhesions
* History of abdominal radiation treatment
* History of pancreatitis within the past 12 months
* History of malabsorption
* Laxative users, except those on stable doses within one (1) month prior to Screening Visit
* History of hepatitis B or C
* History of human immunodeficiency virus (HIV)
* History of cancer within the past five (5) years (except adequately-treated localized basal cell skin cancer or in situ uterine cervical cancer)
* Any other clinically significant disease interfering with the assessments of Gelesis200 (e.g., disease requiring corrective treatment, potentially leading to study discontinuation)
* Abnormal serum thyroid-stimulating hormone (TSH)
* HbA1c >8.5% (>69 mmol/mol)
* Serum low-density lipoprotein (LDL) cholesterol

  -≥160 mg/dL (≥4.15 mmol/L)
* Serum triglycerides ≥350 mg/dL (≥3.96 mmol/L)
* Positive test for drugs of abuse in the urine
* Any relevant biochemical abnormality interfering with the assessments of Gelesis200
* Anti-obesity medications (including herbal preparations) within one (1) month prior to
* Screening Visit
* Systemic corticosteroids within one (1) month prior to Screening Visit
* Thyroid hormones or preparations within one (1) month prior to Screening Visit [except stable dose of replacement therapy for at least two (2) months]
* TSH suppression therapy for thyroid cancer
* Estrogen within one (1) month prior to Screening Visit [except stable dose of replacement therapy or contraceptives for at least one (1) month]
* Any other medication known to cause weight loss or weight gain within one (1) month prior to Screening Visit
* Antidiabetic medications within one (1) month prior to Screening Visit [except stable doses of metformin for at least one (1) month in subjects with Type 2 Diabetes]
* Change in medications treating hypertension within one (1) month prior to Screening Visit
* Change in medications treating dyslipidemia within one (1) month prior to Screening Visit
* Anticipated requirement for use of prohibited concomitant medications
* Any other condition that, in the opinion of the Investigator or Sponsor, would interfere with the subject's ability to participate in the study

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-08-22 (Actual); Primary Completion 2019-11-19 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
The first is placebo-adjusted weight loss of ≥3.0%from baseline to Visit 14 in prediabetic subjects or ≥2.0% in diabetic subjects on Gelesis200. | 26 weeks
  Gelesis is observing if subject loose 3% or more of their body weight as a result of their participating in the study.
weight loss of >5.0% in at least 35% of prediabetic subjects or in at least 25% of diabetic subjects on Gelesis200. | 26 weeks
  Gelesis is observing if pre-diabetic or 25% type 2 diabetic subject loose 5% or more of their body weight as a result of their participating in the study.

SECONDARY OUTCOMES:
statistically significant improvement in HbA1c comparing Gelesis200 to placebo in diabetic subjects | 26 weeks
  Gelesis is observing if subject on Gelesis200 improved their HbA1c better than those on placebo.
improvement in FPG status, post-OGTT plasma glucose status, or post-OGTT plasma glucose AUC in ≥50% of subjects on Gelesis200. | 26 weeks
  Gelesis is observing if greater than 50% of subject on Gelesis200 improved FPG status, post-OGTT plasma glucose status, or post-OGTT plasma glucose AUC.

OTHER OUTCOMES:
Number of TEAE for Gelesis200 similar to placebo or clinically acceptable. | 26 weeks
  Gelesis is continue to observe safety and tolerability profiles on subjects taking Gelesis200.

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Heshmati, MD, Study Director — Gelesis, Inc.
Locations (1):
- University of Copenhagan, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bessesen DH. Update on obesity. J Clin Endocrinol Metab. 2008 Jun;93(6):2027-34. doi: 10.1210/jc.2008-0520. PMID 18539769
- [Background] NCD Risk Factor Collaboration (NCD-RisC). Worldwide trends in diabetes since 1980: a pooled analysis of 751 population-based studies with 4.4 million participants. Lancet. 2016 Apr 9;387(10027):1513-1530. doi: 10.1016/S0140-6736(16)00618-8. Epub 2016 Apr 6. PMID 27061677
- [Background] Pi-Sunyer FX. Medical hazards of obesity. Ann Intern Med. 1993 Oct 1;119(7 Pt 2):655-60. doi: 10.7326/0003-4819-119-7_part_2-199310011-00006. PMID 8363192